CLINICAL TRIAL: NCT01177098
Title: Safety and Efficacy of a New Formulation of Bimatoprost/Timolol Ophthalmic Solution Compared With Bimatoprost/Timolol Ophthalmic Solution in Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 192024-050; 2010-021507-24 (EudraCT Number)
Record Dates: First submitted 2010-08-04; First posted 2010-08-06 (Estimated); Results first posted 2013-03-12 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Bimatoprost; Ganfort

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- bimatoprost/timolol formulation A (Experimental): One drop of bimatoprost/timolol formulation A fixed combination ophthalmic solution administered in each eye every morning for 12 weeks.
  Interventions: Drug: bimatoprost /timolol formulation A fixed combination ophthalmic solution
- bimatoprost/timolol fixed combination ophthalmic solution (Active Comparator): One drop of bimatoprost 0.03%/timolol 0.5% fixed combination ophthalmic solution (Ganfort®) administered in each eye every morning for 12 weeks.
  Interventions: Drug: bimatoprost/timolol fixed combination ophthalmic solution

INTERVENTIONS:
Drug: bimatoprost /timolol formulation A fixed combination ophthalmic solution — One drop of bimatoprost/timolol formulation A fixed combination ophthalmic solution administered in each eye every morning for 12 weeks.
  Arms: bimatoprost/timolol formulation A
Drug: bimatoprost/timolol fixed combination ophthalmic solution — One drop of bimatoprost 0.03%/timolol 0.5% fixed combination ophthalmic solution (Ganfort®) administered in each eye every morning for 12 weeks.
  Other Names: GANFORT®
  Arms: bimatoprost/timolol fixed combination ophthalmic solution

SUMMARY:
This study will evaluate the safety and efficacy of bimatoprost/timolol formulation A ophthalmic solution with Ganfort® (bimatoprost 0.03%/timolol 0.5% ophthalmic solution) once daily for 12 weeks in patients with glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patient has ocular hypertension or glaucoma in both eyes
* Requires IOP-lowering therapy in each eye

Exclusion Criteria:

* Active or recurrent eye disease that would interfere with interpretation of study data in either eye
* History of any eye surgery or laser in either eye within 6 months
* Required chronic use of other eye medications during the study
* Anticipated wearing of contact lenses during the study.
* Intermittent use of oral, intramuscular, or intravenous corticosteroids within 21 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 561 (Actual)
Dates: Start 2010-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (9):
- Artesia, California, United States
- Sydney, New South Wales, Australia
- Brno, Czechia
- Leipzig, Germany
- Budapest, Hungary
- Tel Aviv, Israel
- Saint Petersburg, Russia
- Valencia, Spain
- London, England, United Kingdom

REFERENCES:
- [Derived] Goldberg I, Gil Pina R, Lanzagorta-Aresti A, Schiffman RM, Liu C, Bejanian M. Bimatoprost 0.03%/timolol 0.5% preservative-free ophthalmic solution versus bimatoprost 0.03%/timolol 0.5% ophthalmic solution (Ganfort) for glaucoma or ocular hypertension: a 12-week randomised controlled trial. Br J Ophthalmol. 2014 Jul;98(7):926-31. doi: 10.1136/bjophthalmol-2013-304064. Epub 2014 Mar 25. PMID 24667994

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bimatoprost/Timolol Formulation A | Bimatoprost/Timolol Fixed Combination Ophthalmic Solution
Started | 278 | 283
Completed | 269 | 271
Not Completed | 9 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost/Timolol Formulation A | Bimatoprost/Timolol Fixed Combination Ophthalmic Solution | Total
Number analyzed (Participants) | 278 | 283 | 561
Age, Customized [Number; unit: Participants]
  <45 Years | 12 (10.61) | 13 (10.82) | 25 (10.71)
  45 to 65 Years | 132 | 135 | 267
  >65 Years | 134 | 135 | 269
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 162 | 321
  Male | 119 | 121 | 240

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Worse Eye Intraocular Pressure (IOP) at Each Hour Evaluated at Week 12
Description: Intraocular pressure (IOP) is a measurement of the fluid pressure inside the eye. IOP was evaluated at Baseline and Week 12 at Hour 0, Hour 2 and Hour 8 in the worse eye, defined as the eye with the worse (higher) IOP at baseline. A negative number change from baseline indicates a reduction in IOP (improvement).
Time Frame: Baseline, Week 12
Population: Per-protocol population included randomized participants who did not have a protocol violation that significantly affected the conduct or the results of the trial.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Bimatoprost/Timolol Formulation A | Bimatoprost/Timolol Fixed Combination Ophthalmic Solution
Number analyzed (Participants) | 256 | 260
mm Hg
  Baseline_Hour 0 | 25.41 (2.232) | 25.38 (2.209)
  Baseline_Hour 2 (n=255,260) | 24.79 (2.676) | 24.72 (2.470)
  Baseline_Hour 8 (n=254,259) | 23.88 (3.008) | 23.82 (2.747)
  Change from baseline at Week 12_Hour 0 (n=244,237) | -9.06 (3.216) | -8.72 (3.088)
  Change from baseline at Week 12_Hour 2 (n=235,235) | -8.53 (3.520) | -8.38 (3.297)
  Change from baseline at Week 12_Hour 8 (n=237,234) | -7.98 (3.435) | -7.72 (3.172)

2. Primary Outcome: Average Eye Intraocular Pressure (IOP) at Each Hour Evaluated at Week 2
Description: Intraocular pressure (IOP) is a measurement of the fluid pressure inside the eye. Average eye IOP is the average IOP of both eyes and was evaluated at Week 2 at Hour 0, Hour 2 and Hour 8.
Time Frame: Week 2
Population: Intent-to-treat population included all randomized participants.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Bimatoprost/Timolol Formulation A | Bimatoprost/Timolol Fixed Combination Ophthalmic Solution
Number analyzed (Participants) | 278 | 283
mm Hg
  Week 2_Hour 0 | 16.23 (2.746) | 16.49 (2.887)
  Week 2_Hour 2 | 16.05 (2.877) | 16.23 (2.826)
  Week 2_Hour 8 | 15.49 (2.596) | 15.83 (2.987)

3. Secondary Outcome: Change From Baseline in Worse Eye IOP at Each Hour Evaluated at Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: Intent-to-treat population included all randomized participants.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Bimatoprost/Timolol Formulation A | Bimatoprost/Timolol Fixed Combination Ophthalmic Solution
Number analyzed (Participants) | 278 | 283
mm Hg
  Baseline_Hour 0 | 25.34 (2.233) | 25.30 (2.244)
  Baseline_Hour 2 | 24.71 (2.700) | 24.61 (2.536)
  Baseline_Hour 8 | 23.81 (2.989) | 23.80 (2.795)
  Change from baseline at Week 12_Hour 0 | -8.94 (3.290) | -8.51 (3.253)
  Change from baseline at Week 12_Hour 2 | -8.44 (3.646) | -8.08 (3.504)
  Change from baseline at Week 12_Hour 8 | -7.87 (3.496) | -7.52 (3.362)

4. Secondary Outcome: Change From Baseline in Average Eye IOP at Each Hour Evaluated at Week 12
Description: Intraocular pressure (IOP) is a measurement of the fluid pressure inside the eye. Average eye IOP was evaluated at Baseline and Week 12 at Hour 0, Hour 2 and Hour 8. Average eye IOP is defined as the average of the IOP in both eyes. A negative number change from baseline indicates a reduction in IOP (improvement).
Time Frame: Baseline, Week 12
Population: Intent-to-treat population included all randomized participants.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Bimatoprost/Timolol Formulation A | Bimatoprost/Timolol Fixed Combination Ophthalmic Solution
Number analyzed (Participants) | 278 | 283
mm Hg
  Baseline_Hour 0 | 24.94 (2.116) | 24.86 (2.131)
  Baseline_Hour 2 | 24.29 (2.515) | 24.23 (2.426)
  Baseline_Hour 8 | 23.42 (2.904) | 23.36 (2.703)
  Change from baseline at Week 12_Hour 0 | -8.65 (3.109) | -8.30 (3.009)
  Change from baseline at Week 12_Hour 2 | -8.11 (3.392) | -7.86 (3.413)
  Change from baseline at Week 12_Hour 8 | -7.57 (3.395) | -7.27 (3.226)

5. Primary Outcome: Average Eye Intraocular Pressure (IOP) at Each Hour Evaluated at Week 6
Description: Intraocular pressure (IOP) is a measurement of the fluid pressure inside the eye. Average eye IOP is the average IOP of both eyes and was evaluated at Week 6 at Hour 0, Hour 2 and Hour 8.
Time Frame: Week 6
Population: Intent-to-treat population included all randomized participants.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Bimatoprost/Timolol Formulation A | Bimatoprost/Timolol Fixed Combination Ophthalmic Solution
Number analyzed (Participants) | 278 | 283
mm Hg
  Week 6_Hour 0 | 16.28 (2.754) | 16.31 (2.874)
  Week 6_Hour 2 | 15.90 (2.910) | 16.17 (2.894)
  Week 6_Hour 8 | 15.71 (2.755) | 15.82 (2.926)

6. Primary Outcome: Average Eye Intraocular Pressure (IOP) at Each Hour Evaluated at Week 12
Description: Intraocular pressure (IOP) is a measurement of the fluid pressure inside the eye. Average eye IOP is the average IOP of both eyes and was evaluated at Week 12 at Hour 0, Hour 2 and Hour 8.
Time Frame: Week 12
Population: Intent-to-treat population included all randomized participants.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Bimatoprost/Timolol Formulation A | Bimatoprost/Timolol Fixed Combination Ophthalmic Solution
Number analyzed (Participants) | 278 | 283
mm Hg
  Week 12_Hour 0 | 16.29 (2.783) | 16.56 (2.643)
  Week 12_Hour 2 | 16.18 (2.845) | 16.37 (2.699)
  Week 12_Hour 8 | 15.85 (2.786) | 16.09 (2.714)

ADVERSE EVENTS:
Description: The safety population (all treated participants) was used to calculate the number of participants at risk for Serious Adverse Events and Adverse Events.
Arm/Group | Bimatoprost/Timolol Formulation A | Bimatoprost/Timolol Fixed Combination Ophthalmic Solution
Serious Adverse Events (participants affected / at risk) | 4/278 | 4/282
Other Adverse Events (participants affected / at risk) | 59/278 | 55/282
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost/Timolol Formulation A (N=278) | Bimatoprost/Timolol Fixed Combination Ophthalmic Solution (N=282)
Intermittent claudication (Vascular disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost/Timolol Formulation A (N=278) | Bimatoprost/Timolol Fixed Combination Ophthalmic Solution (N=282)
Conjunctival hyperaemia (Eye disorders) | 59 | 55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.